CLINICAL TRIAL: NCT02464605
Title: An Open-Label, Sequential, Ascending Single-Dose Safety, Tolerability, Pharmacokinetic and Pharmacodynamics Study of an Intravenous Infusion of SEL-037 in Subjects With Elevated Blood Uric Acid Levels
Brief Title: Safety and Pharmacodynamics of SEL-037 (Pegsiticase) in Subjects With Elevated Blood Uric Acid Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Selecta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEL-037/101
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SEL-037 (pegsiticase) (Experimental): Pegylated uricase
  Interventions: Biological: SEL-037 (pegsiticase)

INTERVENTIONS:
Biological: SEL-037 (pegsiticase) — Intravenous infusion of SEL-037

SUMMARY:
This Study will evaluate the safety, pharmacokinetics, pharmacodynamics and immunogenicity of a single intravenous infusion of SEL-037 (pegsiticase), a pegylated uricase, in subjects with elevated blood uric acid levels. Uricase is an enzyme that converts uric acid to the readily soluble allantoin that is then excreted.

DETAILED DESCRIPTION:
This Study will evaluate the safety, pharmacokinetics, pharmacodynamics and immunogenicity of a single intravenous infusion of SEL-037 (pegsiticase), a pegylated uricase, in subjects with elevated blood uric acid levels. Uricase is an enzyme that converts uric acid to the readily soluble allantoin that is then excreted. Cohorts of Subjects will be given a single, ascending dose intravenous infusion of SEL-037 and then monitored for safety, uric acid levels and anti-drug-antibodies (ADAs) to SEL-037 for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ages 21 to 75 inclusive. Female subjects must be of non-childbearing potential;
* Has at the Screening Visit a serum uric acid ≥ 6 mg/dL, with or without a history of gout;
* The use of allopurinol, febuxostat (Uloric®), or probenecid as uric acid-lowering therapy is permissible if dosing has been stable for at least the month prior to the Screening Visit
* Has adequate venous access and able to receive IV therapy;
* Evidence of a personally signed and dated informed consent document indicating that subject has been informed of all pertinent aspects of the study;

Exclusion Criteria:

* Prior exposure to any experimental or marketed uricase;
* History of any allergy to pegylated products,
* Glucose-6-phosphate dehydrogenase deficiency or known catalase deficiency;
* History of hematological or autoimmune disorders, is immunosuppressed or immunocompromised;
* Has participated in a clinical trial within 30 days of the Screening;

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by frequency of drug related adverse events, graded by severity | 30 days
  To assess the safety and tolerability of a single infusion of SEL-037 as assessed by frequency of drug related adverse events, graded by severity

SECONDARY OUTCOMES:
Pharmacokinetics of SEL-037 (AUC) | 30 days
  Measurement of the pharmacokinetics of SEL-037 over 30 days by area under the serum concentration versus time curve (AUC)
Pharmacodynamics of SEL-037 (blood uric acid levels) | 30 days
  Pharmacodynamics of SEL-037 by measurement of blood uric acid levels over 30 days
Immunogenicity of SEL-037 (measurement of anti-drug antibody levels) | 30 days
  Immunogenicity of SEL-037 by measurement of anti-drug antibody levels over 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Altoona Center for Clincal Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas

REFERENCES:
- [Derived] Sands E, Kivitz A, DeHaan W, Leung SS, Johnston L, Kishimoto TK. Tolerogenic nanoparticles mitigate the formation of anti-drug antibodies against pegylated uricase in patients with hyperuricemia. Nat Commun. 2022 Jan 12;13(1):272. doi: 10.1038/s41467-021-27945-7. PMID 35022448